CLINICAL TRIAL: NCT04908670
Title: The Effect of Low-grade Spinal Oscillations Compared to a Pain Neuroscience Education Video on Electroencephalogram (EEG) Brain Activity on Individuals With Chronic Spine Pain: Pilot Study. WITH CHRONIC SPINE PAIN: PILOT STUDY
Brief Title: Comparison of the Effect of Spine Grade I and II Manipulation and a PNE Video on Brainwaves: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Gulf Coast University (Other)
Responsible Party: Principal Investigator, Dr. Rob Sillevis,, Assistant Professor, Florida Gulf Coast University
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 2020-30
Record Dates: First submitted 2021-05-06; First posted 2021-06-01 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Chronic Pain; Manipulation; Psychologic
Keywords: Pain neuroscience education; EEG; Spinal manipulation
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Half of the group was assigned randomly to receive intervention 1 and during the second visit intervention 2. The other half received intervention 2 first followed by intervention 1 on subsequent visit
Who Masked: Participant, Investigator
Masking Description: Participant and clinician providing the manipulation on the spine were blinded to the EEG measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNE group (Active Comparator): 5 minute video :Understanding Pain in less than 5 minutes, and what to do about it! https://www.youtube.com/watch?v=C_3phB93rvI.
  Interventions: Behavioral: Understanding Pain in less than 5 minutes, and what to do about it! https://www.youtube.com/watch?v=C_3phB93rvI; Procedure: PA manipulation
- Manipulation group (Active Comparator): PA grade I-II oscillation on C7, T4 and L4
  Interventions: Behavioral: Understanding Pain in less than 5 minutes, and what to do about it! https://www.youtube.com/watch?v=C_3phB93rvI; Procedure: PA manipulation

INTERVENTIONS:
Behavioral: Understanding Pain in less than 5 minutes, and what to do about it! https://www.youtube.com/watch?v=C_3phB93rvI — Watching pain neuroscience education video
Procedure: PA manipulation — Low grade PA manipulation on the cervical, thoracic and lumbar spine

SUMMARY:
The purpose of this study is to determine the effect of the use of a pain neuroscience educational video instruction on brainwave activity and compare this to the effects of a grade I & II PA spinal oscillations of the spine using EEG in individuals with chronic pain.

DETAILED DESCRIPTION:
This quasi-experimental pilot study compared differences in brainwave activity in subjects with chronic spinal pain following PA spinal oscillations and after viewing a 5-minute pain neuroscience educational video.

In this within subject's design all subjects were given the two interventions on two different days. To prevent the order of the intervention to influence the study results the subjects were randomized into two different groups, A and B. Group A received PA spinal oscillations on their first visit and. Group B's underwent the opposite and watched a pain neuroscience education video on their first visit and received PA spinal oscillations on their first visit. Both sessions and interventions were lead and performed by the Doctor of Physical Therapy student under the direct supervision of the lead physical therapist, who is manually trained and holds a Cranio-Facial Certification. In order to standardize the location of the PA spinal oscillation intervention so brain activity and response can be properly compared, C7, T4 and L4 were identified and marked with a pen prior to any measures. Identification of L4 was achieved by placing hands on the subject's iliac crests with thumbs pointing toward one another. Keeping hands straight and parallel to the floor, thumbs will move medially, landing on L4.25 To identify C7, the subject was taken through cervical extension, where C6 will disappear and C7 remains in place.26 Once C7 was located, the spinous processes were palpated and counted until the level of T4, which was marked. Various factors can affect the reliability of this process, such as subject obesity, therapist experience, and anatomical differences.25 Studies show reliability for this method to be low.25,26 However, these studies, as with most, use a small sample size and only using one palpatory landmark for each level examined.25,26 To standardize variables, the methods above were used in conjunction with palpation of surrounding vertebrae. To measure brain wave activity during this study the 14-lead Emotiv EPOC portable EEG headset was used. Each participant wore the headset throughout the measurement and was in a seated position. After the EEG headset was placed properly and connection with the system had been appropriately established the subjects remained seated in a quiet room for three minutes to accommodate to the room environment before the first EEG measurement. After this, a 1-minute EEG recording was taken. This measurement served as the participant's baseline measurement. Group A subjects then received a grade I & II spinal oscillations of three identified segments (C7, T4, and L4), 1 minute per segment for a total of 3 minutes. Directly following this a second 1-minute EEG recording was taken. On the subsequent visit, group A again underwent the three-minute seated accommodation period with the EEG headset on, followed by a 1 minute baseline EEG measurement prior to watching a 5 minute pain neuroscience educational video Understanding Pain in less than 5 minutes, and what to do about it! https://www.youtube.com/watch?v=C_3phB93rvI. A 1-minute EEG recording was taken during the first minute of the video and again during the last minute of the video. Immediately after watching the pain neuroscience educational video a 1-minute EEG recording was taken. The measurement protocol for group B was the same, but in reversed order. They watched the pain neuroscience educational video at their first visit and the PA spinal oscillations on their next visit.

ELIGIBILITY:
Inclusion Criteria:

Subjects in this study were males and female between the ages of 20 to 65 years with chronic lower back pain (> 3 months). Exclusion Criteria:

Exclusion Criteria:

were not meeting the age requirement having pain less than three months having conditions that would be a contraindication for the grade I-II PA spinal oscillations Those with known neurological conditions making EEG measures unreliable.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2020-08-02 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
EEG power in alpha, delta, gamma, and theta waves | 4- 10 seconds measures of all wave bands in one session measures
  alpha, delta, gamma, and theta waves brain wave measures

CONTACTS AND LOCATIONS:
Locations (1):
- Integrated therapy Practice PC, Merrillville, Indiana, United States

IPD SHARING:
Plan to Share IPD: No